CLINICAL TRIAL: NCT05892913
Title: Treatment of Sympathetic Blockade During Spinal Anesthesia in Cesarian Section Patients With Low-dose, Slow-administered Preemptive Atropine
Brief Title: The Effect of Low-dose Atropine on Sympathetic Blockade in Spinal Cesarean Section Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Akcan AKKAYA Prof. MD., Professor Dr., Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAIBU-Anesthesia-AA-03
Record Dates: First submitted 2023-05-27; First posted 2023-06-07 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Pregnancy; Cesarean Section; Anesthesia, Spinal
Keywords: Pregnancy; Cesarean Section; Anesthesia, Spinal; Atropine; Sympatholytic Effect; Spinal
MeSH Terms: interventions — Atropine; Ephedrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efedrine Group (Active Comparator): For sympathetic blockade (SBP<90) if developed in patients in the ephedrine group, a bolus dose of 5 mg/mL ephedrine would be used and repeated if necessary. In case of development of bradycardia (<65/min) in this group, Atropine 0.5 mg/mL would be planned to be administered and repeated if necessary.
  Interventions: Drug: Ephedrine
- Preemptive Atropine Group (Experimental): In the atropine group, it will planned to administer 0.4 mg/4mL diluted atropine in 20 seconds(10mcg/kg), as a slow bolus as bradycardia would expected (10% reduction in peak heart rate after spinal anesthesia). In this group if SBP<90 despite slow dose atropine administration; it will be planed to give efedrine as bolus of 5 mg/mL. And for bradicardia (HR<65/min) it will be planed to give Atropine 0.5 mg/mL.
  Interventions: Drug: Slow dose preemptive Atropine

INTERVENTIONS:
Drug: Slow dose preemptive Atropine — it will planned to administer 0.4 mg/4mL diluted atropine in 20 seconds(10mcg/kg), as a slow bolus as bradycardia would expected (10% reduction in peak heart rate after spinal anesthesia)
  Other Names: Atropine
  Arms: Preemptive Atropine Group
Drug: Ephedrine — For sympathetic blockade (SBP<90) developed in patients in the ephedrine group, a bolus dose of 5 mg/mL ephedrine was used and repeated if necessary.
  Arms: Efedrine Group

SUMMARY:
The most common side effect in cesarean section surgeries performed under spinal anesthesia is hypotension, which is seen in over 80% and can cause significant morbidity for the mother and fetus. This side effect results from the sympathetic blocking effect, which also causes bradycardia.

A combined approach is supported in the prevention and treatment of hypotension, which recommends adequate fluid support, low-dose spinal anesthesia, and appropriate vasopressor (such as ephedrine, and phenylephrine) and, if bradycardia develops, the use of atropine as a parasympatholytic agent.

In this study, the investigators planned to investigate the possible benefits of preemptive administration of atropine, the dose of which is calculated in proportion to the patient's weight, as soon as a 10% decrease in heart rate is detected, in order to balance the sympathetic blockade due to spinal anesthesia in cesarean section operations.

DETAILED DESCRIPTION:
Our study was approved by the Ethics Committee of Bolu Abant Izzet Baysal University, ASA Ι-ΙΙ, ages 18-40, weight 55-105 kg, height 150-175 cm, with an indication for elective cesarean section, and informed consent will be obtained for the study. Sixty pregnant patients at term scheduled for cesarean delivery under spinal anesthesia will be included.

Those who do not require drug administration with fluid therapy, whose hemodynamic changes are within acceptable range, have systemic disease (Diabetes, COPD, Hypertension), have BMI>34, have a diagnosis of preeclampsia/eclampsia or multiple pregnancy, have pathology in the fetus, have hematological problems such as Rh incompatibility, patients with hypersensitivity to local anesthetics and who are in a position to be a contraindication to regional anesthesia applications will be excluded from the study.

Dexamethasone 4 mg IV for antiemetic purposes was planned for all patients as premedication before the intervention. It was planned to record systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MBP), heart rate (HR), oxygen saturation (SpO2) and respiratory rates by noninvasive method by monitoring the patients with the Mindrey device. In all cases, 2 vascular accesses will be opened with an 18 G (Gauge) intravenous cannula. Intravenous pre-loading was planned for all cases, with 300 cc 0.9% NaCl removed in 15 minutes preoperatively.

Patients will be divided into 2 groups by online randomization method.(Studyrandomizer.com) Fixed dose local anesthetic will be preferred in both groups. After all cases are placed on the operating table and given an anatomical position suitable for spinal anesthesia in a sitting position, skin cleaning will be performed under sterile conditions in the area where the intervention will be performed. Appropriate intervertebral space (L3-L4) will be determined and when the free flow of CSF will be seen after entering the subarachnoid space with a sterile 25-27 G pencil point spinal needle (Egemen/ISTANBUL/TURKEY), 15 mg (2.5 mL) pure (isobaric 0.5% bupivacaine( Marcaine 0.5%/Astra Zeneca/England) ) will be applied. After the application, the patient will placed in the supine position and it will be planned to administer 3 L/min O2 by nasal cannula. After spinal anesthesia, it will planned to start 5 ml/kg/hour 0.9% NaCl solution (Neofleks/Ankara/Turkey) as a maintenance fluid for the patients in both groups during the operation.

In both groups, SBP, DBP, MBP, HR and SpO2 measurements will be recorded at 1, 4, 7, 9, 12, 15, 30, 45, 60, 120 and 240 minutes after the patient is placed left lateral tilt position on the table. After the spinal injection, sensory and motor block levels will be recorded every 3 minutes in the first 15 minutes, and then at the 20th, 25th, 30th, 45th and 60th minutes. It has planned to evaluate the level of sensory block as a dermatome level with the hot-cold test, and motor block by using the Bromage Scale.

The preoperative SBP, DBP, MBP, HR, SpO2 will be recorded before hydration and before spinal anesthesia of the patients will be taken as the baseline value.

For sympathetic blockade (SBP<80) developed in patients in the ephedrine group, a bolus dose of 5 mg/mL ephedrine will be used and repeated if necessary. In case of development of bradycardia (<65/min) in this group, Atropine 0.5 mg/mL will be planned to be administered and repeated if necessary.

In the atropine group, it was planned to administer 0.5 mg/4mL diluted atropine in 20 seconds(10mcg/kg), as a slow bolus as bradycardia would expected (10% reduction in peak heart rate after spinal anesthesia). Also in Atropine group if SBP<80 despite slow dose atropine administration it will be planed to give efedrine. And for bradicardia (HR<65/min) it will be planed to give Atropine 0.5 mg/mL.

The differences between total ephedrine&Atropine consumption, HR,SBP and MBP values in both groups were planned to be the primary outcomes of the study. In addition, findings such as DBP value, nausea and dizziness will also be recorded as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

ASA Ι-ΙΙ Ages 18-40 Weight 55-105 kg Height 150-175 cm

Exclusion Criteria:

Who does not require drug administration with fluid therapy Whose hemodynamic changes are within an acceptable range Diabetes COPD Hypertension BMI>34 Preeclampsia/eclampsia Multiple pregnancies Pathology in the fetus Hematological problems such as Rh incompatibility Hypersensitivity to local anesthetics Contraindications to regional anesthesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Heart rate | 1. minunte after spinal block
  Heart rate
Heart rate | 4. minute after spinal block
  Heart rate
Heart rate | 7. minute after spinal block
  Heart rate
Heart rate | 9. minute after spinal block
  Heart rate
Heart rate | 12. minute after spinal block
  Heart rate
Heart rate | 15. minute after spinal block
  Heart rate
Systolic Blood pressure | 1. minute after spinal block
  Systolic Blood pressure
Systolic Blood pressure | 4. minute after spinal block
  Systolic Blood pressure
Systolic Blood pressure | 7. minute after spinal block
  Systolic Blood pressure
Systolic Blood pressure | 9. minute after spinal block
  Systolic Blood pressure
Systolic Blood pressure | 12. minute after spinal block
  Systolic Blood pressure
Systolic Blood pressure | 15. minute after spinal block
  Systolic Blood pressure
Mean Blood Pressure | 1. minute after spinal block
  Mean Blood Pressure
Mean Blood Pressure | 4. minute after spinal block
  Mean Blood Pressure
Mean Blood Pressure | 7. minute after spinal block
  Mean Blood Pressure
Mean Blood Pressure | 9. minute after spinal block
  Mean Blood Pressure
Mean Blood Pressure | 12. minute after spinal block
  Mean Blood Pressure
Mean Blood Pressure | 15. minute after spinal block
  Mean Blood Pressure
Efedrine Consumption | 1. minute after spinal block
  Efedrine Consumption in the first 15 minutes after the spinal block
Efedrine Consumption | 4. minute after spinal block
  Efedrine Consumption in the first 15 minutes after the spinal block
Efedrine Consumption | 7. minute after spinal block
  Efedrine Consumption in the first 15 minutes after the spinal block
Efedrine Consumption | 9. minute after spinal block
  Efedrine Consumption in the first 15 minutes after the spinal block
Efedrine Consumption | 12. minute after spinal block
  Efedrine Consumption in the first 15 minutes after the spinal block
Efedrine Consumption | 15. minute after spinal block
  Efedrine Consumption in the first 15 minutes after the spinal block
Atropine Consumption | 1. minute after spinal block
  Atropine Consumption in the first 15 minutes after the spinal block
Atropine Consumption | 4. minute after spinal block
  Atropine Consumption in the first 15 minutes after the spinal block
Atropine Consumption | 7. minute after spinal block
  Atropine Consumption in the first 15 minutes after the spinal block
Atropine Consumption | 9. minute after spinal block
  Atropine Consumption in the first 15 minutes after the spinal block
Atropine Consumption | 12. minute after spinal block
  Atropine Consumption in the first 15 minutes after the spinal block
Atropine Consumption | 15. minute after spinal block
  Atropine Consumption in the first 15 minutes after the spinal block

CONTACTS AND LOCATIONS:
Overall Officials: Akcan Akkaya, MD., Principal Investigator — Bolu Abant Izzet Baysal university Medical School, Anesthesiology and Reanimation D.
Locations (1):
- Bolu Abant Izzet Baysal university Medical School, Anesthesiology and Reanimation D., Bolu, Turkey (Türkiye)